CLINICAL TRIAL: NCT00731757
Title: A Phase II, Multi-Center, Open Label Study to Determine the Efficacy of Adalimumab in the Treatment of Cutaneous Sarcoidosis
Brief Title: Efficacy Study of Humira in the Treatment of Cutaneous Sarcoidosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Wright State University (Other)
Collaborators: Stanford University (Other)
Responsible Party: Michael P Heffernan, MD, Wright State University School of Medicine, Department of Dermatology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM 04-36
Record Dates: First submitted 2008-08-06; First posted 2008-08-11 (Estimated); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Sarcoidosis; Cutaneous Sarcoidosis
MeSH Terms: conditions — Sarcoidosis | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Patients being treated with Humira.
  Interventions: Drug: Humira

INTERVENTIONS:
Drug: Humira — 80 mg at week 0, then 40 mg weekly from week 1-week 23.

SUMMARY:
The purpose of this study is to determine the safety and efficacy of Humira in the treatment of cutaneous sarcoidosis.

DETAILED DESCRIPTION:
Sarcoidosis is a multisystem disease. Cutaneous involvement occurs in approximately 25% of patients with lesion morphologies varying widely. There is no universally accepted treatment for sarcoidosis. Systemic agents such as oral corticosteroids are frequently necessary for treatment, but long-term therapy is limited by a multitude of serious adverse effects. Steroid-sparing agents such as methotrexate, azathioprine, anti-malarials, pentoxifylline, allopurinol, and thalidomide have been shown beneficial for select patients, but are limited due to significant toxicities of their own or inconsistencies in efficacy.

Infliximab is a chimeric, monoclonal antibody directed against TNF-α and is currently approved by the US Food and Drug Administration (FDA) to treat rheumatoid arthritis, ankylosing spondylitis, and Crohn's disease. Etanercept is a dimeric fusion protein consisting of the extracellular ligand-binding domain of the human TNF receptor linked to the Fc portion of human IgG1. Etanercept has been approved for the treatment of psoriasis, psoriatic arthritis, rheumatoid arthritis, and juvenile rheumatoid arthritis. Treatment with infliximab and etanercept was generally well tolerated and safe in these reports.

To date, there have been no reports describing the treatment of sarcoidosis with adalimumab. Adalimumab (Humira; Abbott Laboratories, Abbot Park, IL) is a fully human, monoclonal antibody directed against TNF-α and is approved by the US FDA to treat rheumatoid arthritis. Given that adalimumab targets the same cytokine as infliximab and etanercept, one would expect that adalimumab may also be effective in the treatment of sarcoidosis. Treatment with adalimumab is advantageous over infliximab through differences in drug delivery. Infliximab is delivered intravenously in the office. This requires routine office visits and vital sign monitoring by a health care professional.

Adalimumab, on the other hand, is administered subcutaneously once weekly or every other week by the patient at home. Patients can be instructed on proper injection technique during one nurse visit. Additionally, because adalimumab is fully human, patients may be less likely to form antibodies against the medication. Because of the lack of alternative safe, effective treatment for sarcoidosis, a clinical trial to evaluate the efficacy of adalimumab in the treatment of sarcoidosis is warranted.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to give informed consent.
* Subject is willing and able to participate in the study as an outpatient and is willing to comply with study requirements.
* Subject is 18 years of age or older.
* Subject has a diagnosis of cutaneous sarcoidosis for greater than 6 months with a physician global assessment score of at least 4. Diagnosis (based on the recommendations of an expert panel 24) can be made by either:

  * Skin lesions characteristic of sarcoidosis and a biopsy showing granulomas with no evidence of mycobacteria, fungus, or malignancy.
  * A biopsy that does not show granulomas, but the patient has characteristic skin lesions and another clinical feature suggesting sarcoidosis (bilateral hilar adenopathy, erythema nodosum, uveitis, raised ACE level, BAL lymphocytosis (CD4:CD8>3.5), panda/lambda sign on gallium scan)
* If female of childbearing potential, subject will have a negative urine pregnancy test at Screening and Week 0.
* If female, subject will be either post-menopausal for > 1 year, surgically sterile (hysterectomy or bilateral tubal ligation), or practicing one form of birth control (abstinence, oral contraceptive, estrogen patch, implant contraception, injectable contraception, IUD, diaphragm, condom, sponge, spermicides, or vasectomy of partner). Female subjects will continue to use contraception for 6 months following the last infusion.
* Screening laboratory results are within the following parameters:

  * Hemoglobin > 9 g/dL
  * White blood cells > 3.0 x 10 to the 9th power/L, <14.0 x 10 to the 9th power/L (unless on oral corticosteroids and no signs/symptoms of infection)
  * Neutrophils > 1.5 x 10to the 9th power/L
  * Platelets > 100 x 10 to the 9th power/L
  * Lymphocytes > 0.5 x 10 to the 9th power/L
  * Serum creatinine within 1.5 times the upper limit of normal range
  * AST and ALT within 2 times the upper limit of normal range
* Subject has been on a stable dose of antibiotics, thalidomide, antimalarials, oral corticosteroids or other immunosuppressives, such cyclosporine, tacrolimus, azathioprine, methotrexate, or mycophenolate mofetil over the previous 4 weeks.

Exclusion Criteria:

* Subject has evidence of a clinically significant, unstable or poorly controlled medical condition including unstable systemic sarcoidosis.
* Subject has a chest X-ray consistent with an active infection or previous exposure to TB and/or a positive purified protein derivative test at screening (>5 mm).
* Subject has a serious, active or recurrent bacterial, viral, or fungal infection. This includes hepatitis B and C, and HIV.
* Subject has been hospitalized for infection or received IV antibiotics within the previous 2 months prior to baseline.
* Subject has a history of tuberculosis at anytime or close contact with a person with active tuberculosis within the previous 6 months.
* Subject has received a live vaccination within the previous 3 months.
* Subject has a history of a central nervous system disorder/demyelinating disease or symptoms suggestive of multiple sclerosis or optic neuritis.
* Subject has current signs or symptoms or history of systemic lupus erythematosus.
* Subject has been diagnosed with a malignancy within the past 5 years except for successfully treated non-melanoma skin cancer.
* Subject has signs or symptoms suggestive of a possible lymphoproliferative disease.
* Subject has a diagnosis of severe congestive heart failure (Class III or IV NYHA).
* Subject has had a substance abuse problem within the previous 3 years.
* Subject has any dermatologic disease in the target site that may be exacerbated by treatment or interfere with examination.
* Subject has been treated with an anti-TNF biologic immune response modifier, such as infliximab, adalimumab, or etanercept within the past 8 weeks.
* Subject has been treated with topical corticosteroids, tacrolimus, or pimecrolimus within 2 weeks or intralesional corticosteroids within 4 weeks of baseline.
* Subject has been administered an investigational drug in another clinical study within 30 days prior to baseline (or 5 half-lives, whichever is longer).
* Subject has a known allergy to adalimumab.
* Subject is female and is pregnant, is considering becoming pregnant during the study and for 6 months afterwards, or is nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Change in Physician Global Assessment score from baseline to Week 24. | week 0 and week 24.
Change in Physician Target Lesion Assessment score from baseline to Week 24. | Week 0 and week 24.

SECONDARY OUTCOMES:
Number of complete responders, partial responders, minimal responders, and non-responders at Week 24. | Week 0, week 1, week 4 and then every 4 weeks until week 24.
Mean change in Body Surface Area by visit. | Week 0, week 1, week 4 and then every 4 weeks until week 24.
Change in Physician Global Assessment score by visit. | Week 0, week 1, week 4 and then every 4 weeks until week 24.
Change in Physician Target Lesion Assessment score by visit. | Week 0, week 1, week 4 and then every 4 weeks until week 24.
Mean change in the subject's evaluation of severity as measured by a 100 millimeter visual analogue scale by visit. | Week 0, week 1, week 4 and then every 4 weeks until week 24.
Change in dose of antibiotics and immunosuppressives used to treat sarcoid. | Week 0, week 1, week 4 and then every 4 weeks until week 24.

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Heffernan, MD, Principal Investigator — Wright State University
Locations (1):
- Stanford University, Stanford, California, United States